CLINICAL TRIAL: NCT02347332
Title: Phase III Study of IV Vinflunine in Combination With Methotrexate Versus Methotrexate Alone in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck Previously Treated With Platinum-based Chemotherapy
Brief Title: Phase III Study of Vinflunine Plus Methotrexate Versus Methotrexate Alone in Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L00070 IN 309 F0
Record Dates: First submitted 2014-11-18; First posted 2015-01-27 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Recurrent or Metastatic Head and Neck Carcinoma
Keywords: Vinflunin; Vinflunin + Methotrexate; Metastatic Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Recurrence; Squamous Cell Carcinoma of Head and Neck | interventions — vinflunine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vinflunine plus methotrexate (Experimental): vinflunine IV 280 mg/m² Day 1 plus methotrexate IV 30 mg/m² Day 1 and Day 8 every 3 weeks
  Interventions: Drug: Vinflunine
- Methotrexate (Active Comparator): methotrexate IV 40 mg/m² Day 1, 8 and 15 every 3 weeks
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Vinflunine
  Other Names: JAVLOR; VFL
  Arms: Vinflunine plus methotrexate
Drug: Methotrexate
  Other Names: MTX
  Arms: Methotrexate

SUMMARY:
For patients relapsing after platinum-based therapy, few data are available. The current use of cetuximab associated with radiotherapy in localized disease and associated with platinum-based chemotherapy in the first-line setting stresses the need for new therapeutic options at later stages of SCCHN.Vinca-alkaloids demonstrated activity in SCCHN. Vinflunine demonstrated superior antitumour activity to vinorelbine in preclinical animal models. Recent preliminary phase I results of the vinflunine plus methotrexate combination in SCCHN, based on a clinical review, show encouraging antitumour activity and an acceptable safety profile. Therefore the combination of vinflunine and methotrexate appears a promising salvage regimen after platinum failure.

The present study has been designed as a multicenter, randomised phase III study which will compare the combination of IV vinflunine with methotrexate to methotrexate alone in SCCHN patients having failed platinum-based therapy.

DETAILED DESCRIPTION:
This study was designed to compare the OS of VFL plus MTX versus MTX alone in patients with SCCHN who had failed platinum-based chemotherapy.

The trial was designed in accordance with current standards used routinely in oncology phase III trials and used established methods of assessment. The RECIST (version 1.1) and NCI CTCAE (version 3.0) guidelines are internationally recognised methods for assessing efficacy and tolerance, respectively.

The patient population was appropriate for this type of phase III study and included adult patients with recurrent and/or metastatic squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx, who had received prior chemotherapy regimens with documented progression. This population of patients was considered appropriate to meet the study objectives.

Recent preliminary phase I results of the VFL plus MTX combination in SCCHN, reported in a clinical review, showed encouraging antitumour activity and an acceptable safety profile A number of chemotherapy agents have been reported as having single-agent activity in SCCHN. However, reliable evidence of efficacy in the second-line setting is lacking, and there is currently no established standard of care. MTX used alone as the reference regimen at a dose of 40 mg/m2/week can be considered as the best available evidence-based option. Also, other trials using this comparator have demonstrated that it is generally accepted as a reasonable choice, and is often used in general practice.

The efficacy and safety assessments employed in this study are standard measures routinely used in studies of this type

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent and/or metastatic squamous cell carcinoma
* Documented progressive disease after chemotherapy for locoregionally advanced or recurrent/metastatic SCCHN which included a platinum derivative
* Measurable or non measurable disease
* adequate haematological, hepatic and renal functions
* WHO performance status < 1

Exclusion Criteria:

* Nasopharyngeal carcinoma
* History of brain or leptomeningeal involvement
* Albumin level < 35 g/L
* Patients with weight loss ≥ 5% within the last 3 months
* Grade > 2 peripheral neuropathy at study entry
* "Third space" fluids (pleural effusion, ascites, massive edema)
* Prior treatment with vinca-alkaloids and methotrexate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2014-04-25 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2018-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zahida Issiakhem, MD, Study Director — Institut de Recherche Pierre Fabre
Locations (1):
- Institut de Recherche Pierre Fabre, Toulouse, France

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 patients in VFL+MET arrm and 2 patients in MET arm did not receive any treatement. These patients excluded from safety population.
Groups:
- Vinflunine Plus Methotrexate: Vinflunine IV 280 mg/m² day 1 plus methotrexate IV 30 mg/m² Day 1 and Day 8 every 3 weeks
  Vinflunine
- Methotrexate: Methotrexate IV 40 mg/m² days 1, 8 and 15 every 3 weeks
  Methotrexate
Period: Overall Study
Arm/Group | Vinflunine Plus Methotrexate | Methotrexate
Started | 230 | 229
Completed (Were considered as discontinued the 12 patients dead due to various or unknown reasons.) | 0 (6 patients: suicide(1), unknown cause(5 - 4 at home +1 in city hospital).) | 0 (6 patients: unknown cause(2home), PDsuspect(1home+1hosp), sudden death(1home), hypercapnie(1hosp).)
Not Completed | 230 | 229
Not completed — Not treated | 5 | 2
Not completed — Progressive disease | 141 | 159
Not completed — Adverse Event | 50 | 41
Not completed — Death (Unknown, Various reasons) | 6 | 6
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 4 | 3
Not completed — Withdrawal by Subject | 20 | 14
Not completed — Protocol requirement | 1 | 1
Not completed — Switch Post-Trial program | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vinflunine Plus Methotrexate | Methotrexate | Total
Number analyzed (Participants) | 230 | 229 | 459
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 182 | 175 | 357
  >=65 years | 48 | 54 | 102
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 72
  Male | 193 | 194 | 387
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 4 | 3 | 7
  Belarus | 11 | 10 | 21
  Belgium | 4 | 4 | 8
  Brazil | 21 | 15 | 36
  Estonia | 3 | 2 | 5
  France | 31 | 37 | 68
  Germany | 10 | 6 | 16
  Italy | 19 | 19 | 38
  Mexico | 3 | 2 | 5
  Poland | 12 | 11 | 23
  Russia | 58 | 62 | 120
  Slovakia | 2 | 3 | 5
  Spain | 13 | 13 | 26
  Taiwan | 14 | 14 | 28
  Ukraine | 25 | 28 | 53

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival in the ITT Population (Months)
Description: Time from randomization to the date of death or last follow-up. The survival duration of patients still alive, was censored at the date of last contact or last follow-up.
Time Frame: Participants will be followed till death (if they are not lost for follow-up), an expected average of 7.5 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vinflunine Plus Methotrexate | Methotrexate
Number analyzed (Participants) | 230 | 229
Months | 7.1 [5.7 to 8.4] | 6.8 [6.1 to 8.0]
Statistical Analysis 1: Comparison: Vinflunine Plus Methotrexate vs Methotrexate; Test type: Superiority; p = 0.8329, Log Rank — Threshold significance value p<0.05

2. Secondary Outcome: Progression Free Survival
Description: Time measured from the date of randomisation until date of progression or death from any cause (whichever came first)
Time Frame: an expected average of 4 months
Population: ITT
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vinflunine Plus Methotrexate | Methotrexate
Number analyzed (Participants) | 230 | 229
Months | 2.8 [2.6 to 3.3] | 2.8 [2.1 to 3.1]
Statistical Analysis 1: Comparison: Vinflunine Plus Methotrexate vs Methotrexate; Test type: Superiority; p = 0.3576, Log Rank — Threshold significance value p<0.05

3. Secondary Outcome: Objective Response Rate (ORR)
Description: The objective response is defined as the best response designation recorded across all time points from the date of randomisation until disease progression.
Time Frame: 6 weeks
Measure: Median (95% Confidence Interval); unit: Percent of participants
Arm/Group | Vinflunine Plus Methotrexate | Methotrexate
Number analyzed (Participants) | 230 | 229
Percent of participants | 17.8 [13.1 to 23.4] | 14.8 [10.5 to 20.1]
Statistical Analysis 1: Comparison: Vinflunine Plus Methotrexate vs Methotrexate; Test type: Superiority; p = 0.467, Log Rank — Threshold significance value p<0.05

4. Secondary Outcome: Disease Control Rate
Description: Percentage of best overall responses CR, PR and SD in the analysed population
Time Frame: 30 months
Measure: Median (95% Confidence Interval); unit: % patients
Arm/Group | Vinflunine Plus Methotrexate | Methotrexate
Number analyzed (Participants) | 230 | 229
% patients | 50.9 [44.2 to 57.5] | 46.3 [39.7 to 53.0]
Statistical Analysis 1: Comparison: Vinflunine Plus Methotrexate vs Methotrexate; Test type: Superiority; p = 0.243, Log Rank — Threshold significance value p<0.05

5. Secondary Outcome: Duration of Response
Description: Duration of objective response will be measured for responders (CR+PR) from the time for CR or PR until the 1st date of documentation of recurrent or progressive disease or the date of death any cause.
Time Frame: 30 months
Population: ITT
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vinflunine Plus Methotrexate | Methotrexate
Number analyzed (Participants) | 230 | 229
Months | 4.2 [2.5 to 5.6] | 4.2 [2.7 to 5.1]
Statistical Analysis 1: Comparison: Vinflunine Plus Methotrexate vs Methotrexate; Test type: Superiority; p = 0.6289, Log Rank — Threshold significance value p<0.05

ADVERSE EVENTS:
Time Frame: 4 years 6 months 29 days. 5 subjects in the Vinflunine + Methotrexate arm and 2 patients in the Methotrexate arm did not receive any treatment. These patients were thus excluded from the safety population.The safety population consisted of all patients randomized and treated.
Groups:
- Vinflunine Plus Methotrexate: Vinflunine IV 280mg/m2 Day1 plus Methotrexate IV 30mg/m2 on Day 1 and Dy 8 every 3 cycles
  Vinflunine
Arm/Group | Vinflunine Plus Methotrexate | Methotrexate
All-Cause Mortality (participants affected / at risk) | 185/225 | 194/227
Serious Adverse Events (participants affected / at risk) | 106/225 | 81/227
Other Adverse Events (participants affected / at risk) | 211/225 | 213/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vinflunine Plus Methotrexate (N=225) | Methotrexate (N=227)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 16
Tumour Haemorrage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 10
Tumour Necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Neutropenia (Blood and lymphatic system disorders) | 22 | 5
Anaemia (Blood and lymphatic system disorders) | 7 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 1
Leukopenia (Blood and lymphatic system disorders) | 8 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 6
Death (General disorders) | 5 | 6
General Physical Health Deterioration (General disorders) | 6 | 1
Pneumonia (Infections and infestations) | 5 | 5
Sepsis (Infections and infestations) | 8 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vinflunine Plus Methotrexate (N=225) | Methotrexate (N=227)
Weight decreased (Investigations) | 69 (248) | 63 (150)
Creatinine renal clearance decreased (Investigations) | 17 (49) | 10 (28)
Weight increased (Investigations) | 12 (47) | 15 (227)
Alanine aminotransferase increased (Investigations) | 11 (26) | 28 (74)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 (58) | 12 (29)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 16 (16)
Dyspnoea (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (26) | 18 (34)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (32) | 22 (52)
Neutropenia (Blood and lymphatic system disorders) | 89 (219) | 71 (190)
Anaemia (Blood and lymphatic system disorders) | 82 (245) | 56 (147)
Leukopenia (Blood and lymphatic system disorders) | 32 (93) | 38 (102)
Febrile neutropenia (Blood and lymphatic system disorders) | 19 (20) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (31) | 24 (65)
Headache (Nervous system disorders) | 24 (42) | 10 (27)
Asthenia (General disorders) | 62 (181) | 54 (137)
Pyrexia (General disorders) | 26 (35) | 27 (53)
Fatigue (General disorders) | 24 (52) | 27 (53)
Pain (General disorders) | 19 (48) | 17 (55)
Constipation (Gastrointestinal disorders) | 56 (163) | 25 (42)
Stomatitis (Gastrointestinal disorders) | 53 (117) | 64 (158)
Nausea (Gastrointestinal disorders) | 36 (66) | 23 (40)
Vomiting (Gastrointestinal disorders) | 26 (37) | 13 (20)
Diarrhoea (Gastrointestinal disorders) | 23 (34) | 13 (23)
Dysphagia (Gastrointestinal disorders) | 18 (33) | 13 (45)
Abdominal pain (Gastrointestinal disorders) | 16 (18) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 14 (40) | 12 (30)
Decreased appetite (Metabolism and nutrition disorders) | 27 (59) | 23 (45)

LIMITATIONS AND CAVEATS:
Sponsor ended recrutement and decided to limit analysis of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-02-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT02347332/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT02347332/SAP_001.pdf